CLINICAL TRIAL: NCT00202540
Title: Efficacy of 15 mg and 50 mg of S18986 on Cognitive Symptoms in Mild Cognitive Impairment Patients Treated Over a 12-month Oral Administration Period
Brief Title: Efficacy and Safety of S18986 in the Treatment of Mild Cognitive Impairment Patients
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: Institut de Recherches Internationales Servier (Other)
Organization: Servier (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double
Other Study IDs: CL2-18986-009
Record Dates: First submitted 2005-09-12; First posted 2005-09-20 (Estimated); Last update posted 2024-07-25 (Actual); Status verified 2024-07

CONDITIONS: Mild Cognitive Impairment
MeSH Terms: conditions — Cognitive Dysfunction | interventions — S18986-1

INTERVENTIONS:
Drug: S18986

SUMMARY:
The purpose of this study is to demonstrate a long term efficacy of S18986 versus placebo on episodic memory performance in patients with MCI

ELIGIBILITY:
Inclusion Criteria:

* Memory complaint
* Acetylcholinesterase inhibitors stopped at least 3 months before selection

Exclusion Criteria:

* Dementia
* Parkinson's disease
* Vascular disorder
* Depression
* Epilepsy

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2005-06; Primary Completion 2006-03-29 (Actual); Study Completion 2006-03-29 (Actual)

PRIMARY OUTCOMES:
Episodic memory

SECONDARY OUTCOMES:
Other cognitive domains, activities of daily living, global impression of change, MRI, safety.

CONTACTS AND LOCATIONS:
Overall Officials: Bruno Vellas, MD, Study Chair — Hôpital la Grave-Casselardit, Toulouse
Locations (1):
- Hôpital la Grave-Casselardit, Toulouse, France

IPD SHARING:
Plan to Share IPD: Yes
Researchers can ask for a study protocol, patient-level and/or study-level clinical trial data including clinical study reports (CSRs).
  They can ask all interventional clinical studies:
  * submitted for new medicines and new indications approved after 1 January 2014 in the European Economic Area (EEA) or the United States (US).
  * Where Servier or an affiliate are the Marketing Authorization Holders (MAH). The date of the first Marketing Authorization of the new medicine (or the new indication) in one of the EEA Member States will be considered within this scope.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: After Marketing Authorisation in EEA or US if the study is used for the approval.
Access Criteria: Researchers should register on Servier Data Portal and fill in the research proposal form. This form in four parts should be fully documented. The Research Proposal Form will not be reviewed until all mandatory fields are completed.
URL: http://clinicaltrials.servier.com